CLINICAL TRIAL: NCT01277419
Title: German Spondyloarthritis Inception Cohort
Acronym: GESPIC
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); AbbVie (Industry); Amgen (Industry); Centocor, Inc. (Industry); Schering-Plough (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry); Berlin Institute of Health (Other); Novartis (Industry); UCB Pharma (Industry)
Responsible Party: Principal Investigator, Denis Poddubnyy, Prof., Charite University, Berlin, Germany
Other Study IDs: GESPIC
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Ankylosing Spondylitis (AS) / Radiographic Axial SpA (r-axSpA); Non-radiographic Axial Spondyloarthritis (Nr-axSpA); Axial Psoriatic Arthritis (axPsA); Acute Anterior Uveitis (AAU); Crohn Disease (CD); Ulcerative Colitis (UC)
MeSH Terms: conditions — Spondylitis, Ankylosing; Non-Radiographic Axial Spondyloarthritis; Uveitis, Anterior; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (6):
- Ankylosing spondylitis: Ankylosing spondylitis according to the modified New York criteria or with the clinical diagnosis of AS/r-axSpA fulfilling the ASAS Classification Criteria AND the mNY criteria plus having the indiaction for starting a bDMARD therapy according to the treating rheumatologist
- Non-radiographic axial spondyloarthritis: Patients with clinical characteristics of axial SpA but not fulfilling the modified New York criteria for which radiographic sacroiliitis is essential or with the clinical diagnosis of nr-axSpA fulfilling the ASAS Classification Criteria not fulfilling the mNY criteria and the indiaction for starting a bDMARD therapy according to the treating rheumatologist
- Juvenile spondyloarthritis: Patients with juvenile spondyloarthritis (juvenile ankylosing spondylitis, juvenile non-AS-spondyloarthritis).
- Crohn's disease: Patients with Crohn's disease
- Acute anterior uveitis: Patients with acute anterior uveitis
- Axial psoriatic arthritis: Patients with the clinical diagnosis of psoriatic arthritis with axial involvement (sacroiliac joints and/or spine) (axPsA)

SUMMARY:
The German Spondyloarthritis Inception cohort (GESPIC) was started 2000 as a prospective, longitudinal, multicentre, nationwide study in Germany on patients with early SpA including ankylosing spondylitis (AS, also known as radiographic axial spondyloarthritis) and non-radiographic axial SpA. The objectives of GESPIC are to learn about the course of SpA during the very early stage of the disease, to appropriately assess the outcome including radiographic progression of patients after several years of follow-up, to identify outcome predictors, to assess quality of life, function, and costs (direct and indirect costs). GESPIC has been recently expanded to recruit patients with other forms of SpA / conditions associated with SpA: acute anterior uveitis, Crohn's disease as well as with psoriasis / axial psoriatic arthritis.

ELIGIBILITY:
Main inclusion Criteria:

* Patients with definite diagnosis of axial spondyloarthritis or juvenile spondyloarthritis.
* Patients with definite diagnosis of Crohn's disease.
* Patients with definite diagnosis of acute anterior uveitis.
* Patients with definite diagnosis of psoriatic arthritis with axial involvement.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients included in GESPIC are required to have a definite clinical diagnosis of axial SpA / juvenile SpA (currently only adult patients with radiographic axial SpA = ankylosing spondylitis - AS are recruited) or a definite diagnosis of Crohn's disease or a definite diagnosis of acute anterior uveitis or a definite diagnosis of psoriatic arthritis with axial involvement.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2000-07; Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Sieper, Prof. Dr., Study Chair — Charite University, Berlin, Germany; Martin Rudwaleit, Prof. Dr., Study Chair — Charite University, Berlin, Germany; Denis Poddubnyy, Prof. Dr., Study Chair — Charite University, Berlin, Germany; Fabian Proft, MD, Study Chair — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Result] Rudwaleit M, Haibel H, Baraliakos X, Listing J, Marker-Hermann E, Zeidler H, Braun J, Sieper J. The early disease stage in axial spondylarthritis: results from the German Spondyloarthritis Inception Cohort. Arthritis Rheum. 2009 Mar;60(3):717-27. doi: 10.1002/art.24483. PMID 19248087
- [Result] Poddubnyy DA, Rudwaleit M, Listing J, Braun J, Sieper J. Comparison of a high sensitivity and standard C reactive protein measurement in patients with ankylosing spondylitis and non-radiographic axial spondyloarthritis. Ann Rheum Dis. 2010 Jul;69(7):1338-41. doi: 10.1136/ard.2009.120139. Epub 2010 May 24. PMID 20498207
- [Result] Poddubnyy D, Rudwaleit M, Haibel H, Listing J, Marker-Hermann E, Zeidler H, Braun J, Sieper J. Rates and predictors of radiographic sacroiliitis progression over 2 years in patients with axial spondyloarthritis. Ann Rheum Dis. 2011 Aug;70(8):1369-74. doi: 10.1136/ard.2010.145995. Epub 2011 May 27. PMID 21622969
- [Result] Poddubnyy DA, Marker-Hermann E, Kaluza-Schilling W, Zeidler H, Braun J, Listing J, Sieper J, Rudwaleit M. Relation of HLA-B27, tumor necrosis factor-alpha promoter gene polymorphisms, and T cell cytokine production in ankylosing spondylitis -- a comprehensive genotype-phenotype analysis from an observational cohort. J Rheumatol. 2011 Nov;38(11):2436-41. doi: 10.3899/jrheum.110130. Epub 2011 Sep 1. PMID 21885496
- [Result] Heiland GR, Appel H, Poddubnyy D, Zwerina J, Hueber A, Haibel H, Baraliakos X, Listing J, Rudwaleit M, Schett G, Sieper J. High level of functional dickkopf-1 predicts protection from syndesmophyte formation in patients with ankylosing spondylitis. Ann Rheum Dis. 2012 Apr;71(4):572-4. doi: 10.1136/annrheumdis-2011-200216. Epub 2011 Dec 20. PMID 22186710
- [Result] Poddubnyy D, Rudwaleit M, Haibel H, Listing J, Marker-Hermann E, Zeidler H, Braun J, Sieper J. Effect of non-steroidal anti-inflammatory drugs on radiographic spinal progression in patients with axial spondyloarthritis: results from the German Spondyloarthritis Inception Cohort. Ann Rheum Dis. 2012 Oct;71(10):1616-22. doi: 10.1136/annrheumdis-2011-201252. Epub 2012 Mar 29. PMID 22459541
- [Result] Poddubnyy D, Haibel H, Listing J, Marker-Hermann E, Zeidler H, Braun J, Sieper J, Rudwaleit M. Cigarette smoking has a dose-dependent impact on progression of structural damage in the spine in patients with axial spondyloarthritis: results from the GErman SPondyloarthritis Inception Cohort (GESPIC). Ann Rheum Dis. 2013 Aug;72(8):1430-2. doi: 10.1136/annrheumdis-2012-203148. Epub 2013 Apr 26. No abstract available. PMID 23625981
- [Result] Poddubnyy D, Conrad K, Haibel H, Syrbe U, Appel H, Braun J, Rudwaleit M, Sieper J. Elevated serum level of the vascular endothelial growth factor predicts radiographic spinal progression in patients with axial spondyloarthritis. Ann Rheum Dis. 2014 Dec;73(12):2137-43. doi: 10.1136/annrheumdis-2013-203824. Epub 2013 Aug 16. PMID 23956246
- [Result] Turina MC, Sieper J, Yeremenko N, Conrad K, Haibel H, Rudwaleit M, Baeten D, Poddubnyy D. Calprotectin serum level is an independent marker for radiographic spinal progression in axial spondyloarthritis. Ann Rheum Dis. 2014 Sep;73(9):1746-8. doi: 10.1136/annrheumdis-2014-205506. Epub 2014 May 20. No abstract available. PMID 24845387
- [Result] Syrbe U, Callhoff J, Conrad K, Poddubnyy D, Haibel H, Junker S, Frommer KW, Muller-Ladner U, Neumann E, Sieper J. Serum adipokine levels in patients with ankylosing spondylitis and their relationship to clinical parameters and radiographic spinal progression. Arthritis Rheumatol. 2015 Mar;67(3):678-85. doi: 10.1002/art.38968. PMID 25417763
- [Result] Poddubnyy D, Haibel H, Braun J, Rudwaleit M, Sieper J. Brief Report: Clinical Course Over Two Years in Patients With Early Nonradiographic Axial Spondyloarthritis and Patients With Ankylosing Spondylitis Not Treated With Tumor Necrosis Factor Blockers: Results From the German Spondyloarthritis Inception Cohort. Arthritis Rheumatol. 2015 Sep;67(9):2369-75. doi: 10.1002/art.39225. PMID 26017497
- [Result] Poddubnyy D, Protopopov M, Haibel H, Braun J, Rudwaleit M, Sieper J. High disease activity according to the Ankylosing Spondylitis Disease Activity Score is associated with accelerated radiographic spinal progression in patients with early axial spondyloarthritis: results from the GErman SPondyloarthritis Inception Cohort. Ann Rheum Dis. 2016 Dec;75(12):2114-2118. doi: 10.1136/annrheumdis-2016-209209. Epub 2016 Apr 28. PMID 27125522
- [Result] Protopopov M, Sieper J, Haibel H, Listing J, Rudwaleit M, Poddubnyy D. Relevance of structural damage in the sacroiliac joints for the functional status and spinal mobility in patients with axial spondyloarthritis: results from the German Spondyloarthritis Inception Cohort. Arthritis Res Ther. 2017 Oct 24;19(1):240. doi: 10.1186/s13075-017-1453-3. PMID 29065931
- [Result] Poddubnyy D, Listing J, Haibel H, Knuppel S, Rudwaleit M, Sieper J. Functional relevance of radiographic spinal progression in axial spondyloarthritis: results from the GErman SPondyloarthritis Inception Cohort. Rheumatology (Oxford). 2018 Apr 1;57(4):703-711. doi: 10.1093/rheumatology/kex475. PMID 29373733
- [Result] Boel A, Molto A, van der Heijde D, Ciurea A, Dougados M, Gensler LS, Santos MJ, De Miguel E, Poddubnyy D, Rudwaleit M, van Tubergen A, van Gaalen FA, Ramiro S. Do patients with axial spondyloarthritis with radiographic sacroiliitis fulfil both the modified New York criteria and the ASAS axial spondyloarthritis criteria? Results from eight cohorts. Ann Rheum Dis. 2019 Nov;78(11):1545-1549. doi: 10.1136/annrheumdis-2019-215707. Epub 2019 Jul 30. PMID 31362994
- [Result] Llop M, Rios Rodriguez V, Redeker I, Sieper J, Haibel H, Rudwaleit M, Poddubnyy D. Incorporation of the anteroposterior lumbar radiographs in the modified Stoke Ankylosing Spondylitis Spine Score improves detection of radiographic spinal progression in axial spondyloarthritis. Arthritis Res Ther. 2019 May 24;21(1):126. doi: 10.1186/s13075-019-1913-z. PMID 31126334
- [Result] de Winter JJ, Blijdorp IC, de Jong HM, Sauter J, Schmidt AH, van Gaalen FA, van der Heijde D, Poddubnyy D, Yeremenko NG, van de Sande MG, Baeten DL. HLA-C*07 in axial spondyloarthritis: data from the German Spondyloarthritis Inception Cohort and the Spondyloarthritis Caught Early cohort. Genes Immun. 2019 Nov;20(8):671-677. doi: 10.1038/s41435-019-0061-4. Epub 2019 Feb 26. PMID 30809016
- [Derived] Weiss A, Minden K, Listing J, Foeldvari I, Sieper J, Rudwaleit M. Course of patients with juvenile spondyloarthritis during 4 years of observation, juvenile part of GESPIC. RMD Open. 2017 Mar 21;3(1):e000366. doi: 10.1136/rmdopen-2016-000366. eCollection 2017. PMID 28405472
- See also: Coordinating study center: Department of rheumatology, Charité - Campus Benjamin Franklin — https://rheuma.charite.de